CLINICAL TRIAL: NCT04194671
Title: A Single-center, Randomized, Placebo-controlled, Patient-blinded Study of Mesenchymal Stem Cells Therapy in Subjects With Severe Acute Kidney Injury Receiving Routine Therapy
Brief Title: Clinical Trial of Mesenchymal Stem Cells in the Treatment of Severe Acute Kidney Injury
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiangmei, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSC-001
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Acute Kidney Injury; Mesenchymal Stem Cells
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cells cohort (Experimental)
  Interventions: Biological: Mesenchymal stem cells
- Saline cohort (Placebo Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Mesenchymal stem cells — In experimental group, patients receive standard treatment and allogeneic human umbilical cord derived-mesenchymal stem cells (MSCs) is administered via intravenous infusion on day 0 and day 7
  Arms: Mesenchymal stem cells cohort
Other: Saline — In placebo control group, patients receive standard treatment and saline is administered via intravenous infusion on day 0 and day 7
  Arms: Saline cohort

SUMMARY:
Acute kidney injury(AKI) is a common, severe emergency case in clinics,especially severe AKI ,which is associated with higher morbidity and mortality. Effect of routine therapy is limited and mesenchymal stem cells (MSC)are considered a new therapy for treating severe acute kidney injury. Patients will be randomized to receive intravenous infusion of MSC, or placebo control. This trial is to investigate whether MSC can improve renal recovery and mortality of patients with AKI.

ELIGIBILITY:
Inclusion Criteria:

* Have severe AKI defined as more than two-fold increase serum creatinine level compared with baseline within 48 hours and/or urinary output consistently<0.5 ml/kg/h over 12 hours
* Age between 18 and 65 years
* Willing or having a legally acceptable representative to give a written informed consent
* Able to comply with visit schedule and study procedures including post-hospitalization discharge follow-up

Exclusion Criteria:

* AKI due to post-renal outflow obstruction,glomerulonephritis,lupus nephritis, antineutrophil cytoplasmic antibody (ANCA) related nephritis, antiglomerular basement membrane disease, cryoglobulinemia, thrombotic microangiopathy, and AKI caused by purpura nephritis
* Pregnant or lactating woman
* Allergic person
* Organ transplant or hematopoietic stem cell transplant
* Patients with malignant tumors or those with a history of cancer
* Life expectancy is less than 3 months
* Known end-stage liver disease
* Uncontrollable infection
* Patients younger than 65 years old ,whose estimated glomerular filtration rate (eGFR) were less than 60
* Severe pulmonary dysfunction
* Severe cardiac dysfunction,left ventricular ejection fraction is less than 40%, or severe arrhythmia patients
* Hemodynamically unstable patients
* Organ failure affecting more than 2 non-renal organs
* Acute or chronic vasculitis of any cause
* History of chronic systemic infection of any cause
* The investigators believe that subjects may need to gradually increase the dose of vasopressor to achieve and / or maintain hemodynamic stability
* Systemic immunosuppressive therapy that has not been stabilized for greater than 4 months, or in the case of chronic corticosteroid therapy, a dose of >15 mg/day of prednisone or the equivalent within the past 30 days
* Platelet count <25,000/uL or other severe hematologic abnormalities, causing the subject to be at risk of death
* Patients need mechanical ventilation
* Participate in other clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference in the renal function between the two groups (MSC treatment group vs placebo control group) within 28 days after receiving MSC/ placebo treatment | within 28 days after receiving MSC/ placebo treatment
  Compare the creatinine concentration between the two groups (MSC treatment group vs placebo control group) at 28 days after receiving MSC/ placebo treatment.

SECONDARY OUTCOMES:
Overall survival within 28 days after receiving MSC/ placebo treatment | 28 days
  Compare the overall survival rate between the two groups (MSC treatment group vs placebo control group) at 28 days after receiving MSC/ placebo treatment.
Overall survival within 3 months after receiving MSC/ placebo treatment | 3 months
  Compare the overall survival rate between the two groups (MSC treatment group vs placebo control group) at month 3 after receiving MSC/ placebo treatment.
Renal replacement therapy (RRT) dependent within 3 months after receiving MSC/ placebo treatment | 3 months
  Compare the rate of renal replacement therapy (RRT) dependence between the two groups (MSC treatment group vs placebo control group) at month 3 after receiving MSC/ placebo treatment.
Complete renal recovery within 3 months after receiving MSC/ placebo treatment | 3 months
  Compare the rate of complete renal recovery between the two groups (MSC treatment group vs placebo control group) at month 3 after receiving MSC/placebo treatment. We considered complete recovery as alive, free of RRT, and the SCR decreased to no more than 1.5 times of the baseline level.
Partial renal recovery within 3 months after receiving MSC/ placebo treatment | 3 months
  Compare the rate of partial renal recovery between the two groups (MSC treatment group vs placebo control group) at month 3 after receiving MSC/placebo treatment. Partial recovery refers to survival, free of RRT, and the SCR 1.5 times higher than the baseline level of creatinine.
ICU and hospitalization duration of stay among all AKI patients within 3 months after receiving MSC/ placebo treatment | 3 months
  Compare the days in ICU and hospital between the two groups (MSC treatment group vs placebo control group) at month 3 after receiving MSC/placebo treatment.
Adverse events within 3 months after receiving MSC/ placebo treatment | 3 months
  Compare the rate of adverse events between the two groups (MSC treatment group vs placebo control group) at month 3 after receiving MSC/placebo treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Data will be available beginning immediately following publication and ending 36 months following article publication.

REFERENCES:
- [Derived] Yang Y, Gao J, Wang S, Wang W, Zhu FL, Wang X, Liang S, Feng Z, Lin S, Zhang L, Chen X, Cai G. Efficacy of umbilical cord mesenchymal stem cell transfusion for the treatment of severe AKI: a protocol for a randomised controlled trial. BMJ Open. 2022 Feb 21;12(2):e047622. doi: 10.1136/bmjopen-2020-047622. PMID 35190406